CLINICAL TRIAL: NCT04899492
Title: Pilot Study in Cancer Patients Scheduled for Surgery Evaluating Different Smoking Cessation Protocols : Nicotine Replacement, Motivational Interviewing (MI), Cognitive Behavioural Therapy (CBT) or Hypnotherapy
Brief Title: Evaluation of Different Smoking Cessation Protocols: Nicotine Replacement, Motivational Interviewing (MI), Cognitive Behavioural Therapy (CBT) or Hypnotherapy in Cancer Patients Scheduled for Surgery
Acronym: RESPIRE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of patient enrolment
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2020-14
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Gynecologic Cancer; Digestive Cancer; Melanoma
Keywords: Smoking Cessation; Motivational Interviewing (MI); Cognitive Behavioural Therapy (CBT); Hypnotherapy; Nicotine Replacement Therapy (NRT); Surgery; Surgery complications; longitudinal cohort
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms; Melanoma; Smoking Cessation | interventions — Motivational Interviewing; Cognitive Behavioral Therapy; Hypnosis; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: pilot study, monocentric, prospective, randomization according to Zelen's design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1:Nicotine Replacement Therapy (NRT) (Active Comparator): Patients enrolled in group 1 will receive a Nicotine Replacement Therapy (NRT) from the study entry to end of study
  Interventions: Drug: Nicotine Replacement Therapy (NRT)
- Group 2:Motivational Interviewing (MI) (Experimental): Patients enrolled in group 2 will receive a Nicotine Replacement Therapy (NRT) from the study entry to end of study and 1 to 3 Motivational Interviewing (MI) after randomization
  Interventions: Behavioral: Motivational Interviewing (MI); Drug: Nicotine Replacement Therapy (NRT)
- Group 3:Cognitive Behavioural Therapy (CBT) (Experimental): Patients enrolled in group 3 will receive a Nicotine Replacement Therapy (NRT) from the study entry to end of study and 1 to 3 Motivational Interviewing (MI) after randomization and 6 sessions of CBT after Motivational Interviewing up to 6 months after
  Interventions: Behavioral: Motivational Interviewing (MI); Behavioral: Cognitive Behavioural Therapy (CBT); Drug: Nicotine Replacement Therapy (NRT)
- Group 4: Hypnotherapy (Experimental): Patients enrolled in group 4 will receive a Nicotine Replacement Therapy (NRT) from the study entry to end of study and 1 to 3 Motivational Interviewing (MI) after randomization and about 3 sessions of hypnotherapy up to 6 months after
  Interventions: Behavioral: Motivational Interviewing (MI); Behavioral: Hypnotherapy; Drug: Nicotine Replacement Therapy (NRT)

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — 1 to 3 Motivational Interviewing (MI) should be performed after randomization by a psychotherapist
  Arms: Group 2:Motivational Interviewing (MI); Group 3:Cognitive Behavioural Therapy (CBT); Group 4: Hypnotherapy
Behavioral: Cognitive Behavioural Therapy (CBT) — 6 Cognitive Behavioural Therapy (CBT) sessions should be performed after motivational interviewing up to 6 months by a psychotherapist
  Arms: Group 3:Cognitive Behavioural Therapy (CBT)
Behavioral: Hypnotherapy — About 3 Hypnotherapy sessions should be performed after motivational interviewing up to 6 months by a hypnotherapist
  Arms: Group 4: Hypnotherapy
Drug: Nicotine Replacement Therapy (NRT) — All patients will receive Nicotine Replacement Therapy (NRT) from randomization up to 6 months

SUMMARY:
This trial offers support and assistance to patients wishing to quit smoking in order to increase the success rate of smoking cessation and all the benefits associated with it. Patients will be monitored by a tobacco specialist and will be able to benefit from one or more therapies complementary to Nicotine Replacement Therapy (NRT): Motivational Interviewing (MI), Cognitive Behavioural Therapy (CBT) or Hypnotherapy.

DETAILED DESCRIPTION:
The study RESPIRE is aiming to identify some interventions to be proposed as part of a smoking cessation programme for smokers with cancer requiring surgical treatment and wishing to stop smoking. We aim to compare different smoking cessation methods in addition to the currently recommended treatments: Nicotine Replacement Therapy (NRT). These procedures are: Cognitive Behavioural Therapy (CBT), Motivational Interviewing (MI) or hypnotherapy in order to improve the success rate of smoking cessation in this specific population.

All patients wishing to be supported to stop smoking will be randomized and will be followed by a tobacco specialist before and after surgery. They will receive NRT for 12 months.

Smoking assessment, exhaled CO measurement, questionnaires will be completed regularly to assess depression, anxiety and quality of life during the 12 months.

Patients randomized in group 2 will receive 1 to 3 MI. Patients randomized in group 3 will receive 1 to 3 MI and 6 CBT sessions by a psychotherapist.

Patients randomized in group 4 will receive 1 to 3 MI and at least 3 sessions oh hypnotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Smoking patient: daily tobacco consumption.
* Patient with cancer requiring surgical treatment (breast cancer, digestive cancer, gynecological).
* Patient wishing to quit smoking.
* Fagerström > 3.
* Patient has valid health insurance
* Information and agreement of the patient to participate in the longitudinal cohort.
* Signing of specific informed consent for patients in groups 1 to 4 before any study-related intervention.
* Person able to speak, read and understand French.

Exclusion Criteria:

* Patient not receiving surgical treatment.
* Refusal to participate in the longitudinal cohort study.
* Pregnant or likely to be pregnant or nursing patient.
* Persons deprived of their liberty, under a measure of safeguard of justice, under guardianship or placed under the authority of a guardian
* disability to undergo the medical follow-up of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Testing the feasibility of smoking cessation interventions evaluated in French cancer patients undergoing surgery | 12 months
  Number of patients who completed all planned sessions out of the total number of patients randomised to each group

SECONDARY OUTCOMES:
Evaluate the efficacy of the following interventions for smoking cessation in French cancer patients: MI, CBT and Hypnotherapy, combined with nicotine replacement therapy | 12 months
  Percentage of patients with an exhaled Carbone Monoxide (CO) measurement < 10 ppm at study visits.
Evaluate the efficacy of the following interventions for smoking cessation in French cancer patients: MI, CBT and Hypnotherapy, combined with nicotine replacement therapy | 12 months
  Percentage of patients reporting no smoking during the last 7 days before the visit.
Evaluate the efficacy of the different interventions in reducing tobacco consumption | 12 months
  Number of cigarettes smoked per day from baseline
Evaluate the efficacy of the different interventions in terms of continued abstinence since surgery | 12 months
  Percentage of patients reporting no smoking since surgery
Evaluate the reduction in side effects of oncological treatments after smoking cessation | 3 month
  Report all Grade > 1 side effects of oncology treatments up to 3 months after the end of treatment or the end of the study
Estimate the decrease in surgical complications | 1 month
  Report all surgical complications (Grade > 1 according to Clavien Dindo classification) up to 1 month after surgery
Evaluate the efficacy of interventions on patient depression and anxiety | 12 months
  Patient Depression and anxiety will be evaluated by using the Hospital Anxiety and Depression Scale (HADS)
Evaluate the efficacy of interventions on patient quality of life | 12 months
  Patient quality of life will be evaluated by using the Quality of Life Questionnaire (QLQ-C30)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancerologie de l'Ouest (ICO), Saint-Herblain, France